CLINICAL TRIAL: NCT05952661
Title: Minimal Residual Disease Guided Radical Chemoradiotherapy Combined With Immunotherapy After Neoadjuvant Immunochemotherapy Followed by Adjuvant Immunotherapy for Esophageal Squamous Cell Cancer
Brief Title: Minimally Residual of Esophageal Cancer 001
Acronym: ECMRD-001
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ECMRD-001
Record Dates: First submitted 2023-06-20; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Carcinoma; Minimal Residual Disease
Keywords: circulating tumor DNA; ctDNA; minimal residual disease; MRD; esophageal cancer; esophageal carcinoma; neoadjuvant immunochemotherapy; chemoradiotherapy; adjuvant immunotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The specimen collection time points were divided into MRD-related blood collections, MRD-related tissue collection, T-cell immunohistobank-related blood collections, and T-cell immunohistobank-related tissue collection before, during, and after treatment and follow-up. The investigators will test circulating tumor DNA (ct-DNA) based minimal residual disease (MRD) indicators for research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This trial aims to assess changes in minimal residual disease (MRD) status before and after radical concurrent chemoradiotherapy combined with immunotherapy and adjuvant immunotherapy after neoadjuvant immunochemotherapy in patients with inoperable stage II-III esophageal squamous cell cancer (ESCC), and correlate with the efficacy of adjuvant immunotherapy.

DETAILED DESCRIPTION:
Presence of circulating tumor DNA (ctDNA) is indicative for minimal residual disease (MRD) and has high predictive value for efficacy and tumor recurrence. Concurrent chemoradiotherapy becomes the standard of care for unresectable, locally advanced esophageal squamous cell cancer, and the addition of immunotherapy to radiotherapy has been shown to increase efficacy without increasing side effects. The ECMRD-001 trial aims to assess changes in MRD status before and after radical concurrent chemoradiotherapy combined with immunotherapy and adjuvant immunotherapy after neoadjuvant immunochemotherapy in patients with inoperable stage II-III esophageal squamous cell cancer (ESCC). The specimen collection time points were divided into MRD-related blood collections, MRD-related tissue collection, T-cell immunohistobank-related blood collections, and T-cell immunohistobank-related tissue collection before, during, and after treatment and follow-up. Primary endpoint is the relationship between MRD status at different time points and treatment efficacy. Secondary endpoints include the relationship between MRD status and immune microenvironment, radiotherapy dose, and tumor recurrence. Exploratory endpoint is to investigate ctDNA mutations in ESCC patients receiving adjuvant immunotherapy. To the investigators' knowledge, the ECMRD-001 study is the first clinical trial to investigate ctDNA-based MRD guided strategies in stage II-III ESCC patients who receive radical chemoradiotherapy combined with immunotherapy after neoadjuvant immunochemotherapy followed by adjuvant immunotherapy. After our research it may be possible to confirm that ctDNA-based MRD may be a predictive marker for the efficacy and tumor recurrence of inoperable ESCC patients; elevated ctDNA-MRD may predict tumor recurrence earlier than imaging; ctDNA-based MRD analysis and ctDNA-based MRD guided diagnosis and treatment may be implemented into clinical practice to improve efficacy and reduce tumor recurrence of inoperable stage II-III ESCC.

ELIGIBILITY:
Inclusion Criteria:

1. age: 18 - 75 years
2. gender: both sexes, as balanced as possible
3. patients with clinically confirmed TNM 8th stage II-III ESCC by histopathology and are not suitable for surgery
4. patients receive neoadjuvant immunochemotherapy, followed by radical CCRT combined with immunotherapy and finally adjuvant immunotherapy
5. Eastern Cooperative Oncology Group (ECOG) score: 0-1
6. the functional condition of the organ meets the following requirements- haematological indicators: absolute neutrophil count ≥ 1.5 * 109/L, platelet count ≥ 100 * 109/L, haemoglobin count≥ 9 g/dL; good coagulation: platelet count ≥ 100 x 109/L. Liver: total bilirubin ≤ 2 times the upper limit of normal, ghrelin and ghrelin ≤ 2.5 times the upper limit of normal. Renal: creatinine ≤ 1.5 times the upper limit of normal, or creatinine clearance ≥ 60 mL/min (calculated by the Cockcroft-Gault formula)
7. women of childbearing age must have a urine pregnancy test with a negative result within 7 days prior to starting treatment
8. patients understand and voluntarily sign the informed consent form

Exclusion Criteria:

* (1) patients have been diagnosed or treated for another malignancy within 5 years prior to the start of this study (2) adenocarcinoma, mixed adenosquamous or other pathological types of esophageal cancer (3) any unstable systemic disease, including: active infection, uncontrolled hypertension, unstable angina, angina pectoris starting within the last 3 months, congestive heart failure (≥ New York Heart Association [NYHA] class II), myocardial infarction (6 months prior to enrollment), severe arrhythmia requiring medication, liver, kidney or metabolic disease (4) with known or suspected active autoimmune disease (5) previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or any other antibodies or drugs that specifically target T-cell co-stimulation or checkpoint pathways (6) known history of testing positive for human immunodeficiency virus (HIV) or known to have acquired immunodeficiency syndrome (AIDS) (7) female patients who are pregnant or breastfeeding (8) other conditions deemed unsuitable for enrolment by the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal squamous cell cancer patients who receive radical chemoradiotherapy combined with immunotherapy after neoadjuvant immunochemotherapy followed by adjuvant immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlations of minimal residual disease (MRD) and efficacy | 2023/2/22-2027/12/31
  The changes in MRD status before and after radical CCRT combined with immunotherapy and adjuvant immunochemotherapy in patients with inoperable resectable stage II-III ESCC, correlating with the efficacy of adjuvant immunotherapy

SECONDARY OUTCOMES:
The differences in the efficacy of neoadjuvant immunochemotherapy in patients with positive versus negative blood MRD prior to radical concurrent chemoradiotherapy (CCRT) combined with immunotherapy following neoadjuvant immunochemotherapy | 2023/2/22-2027/12/31
  Differences in overall survival (OS) and progression-free survival (PFS) between MRD positive and negative patients after neoadjuvant immunochemotherapy. OS is defined as time from start of treatment to death (from any cause). PFS is defined as the time between the start of treatment and the onset of (any aspect of) tumor progression or death (from any cause).
The differences in the immune microenvironment in patients with different efficacy responses after radical CCRT combined with immunotherapy | 2023/2/22-2027/12/31
  MRD status and T-lymphocyte differences across efficacy responses after receiving radical CCRT combined with immunotherapy. Therapeutic response is evaluated according to immune-related response evaluation criteria in solid tumors (irRECIST).
The differences in MRD status between radiation doses of 50Gy and 60Gy, and the correlation with patient prognosis | 2023/2/22-2027/12/31
  The differences in MRD status between radiation doses of 50Gy and 60Gy, and the correlation with patient prognosis.
The association between serial changes in MRD status and the efficacy of adjuvant immunotherapy | 2023/2/22-2027/12/31
  The association between serial changes in MRD status and the efficacy of adjuvant immunotherapy. Therapeutic response is evaluated according to immune-related response evaluation criteria in solid tumors (irRECIST).
The timing of MRD advance warning of recurrence in patients ahead of imaging cues | 2023/2/22-2027/12/31
  The timing of MRD advance warning of recurrence in patients ahead of imaging cues

OTHER OUTCOMES:
ctDNA mutation profiles in ESCC patients undergoing adjuvant immunotherapy. | 2023/2/22-2027/12/31
  High-frequency mutated genes in the ESCC patients undergoing adjuvant immunotherapy and the corresponding mutation frequency (percentage of samples with mutations out of all samples).

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Shen, PhD, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Wang H, Zhang X, Zhao X, Song C, Deng W, Shen W. Minimal residual disease guided radical chemoradiotherapy combined with immunotherapy after neoadjuvant immunochemotherapy followed by adjuvant immunotherapy for esophageal squamous cell cancer (ECMRD-001): a study protocol for a prospective cohort study. Front Immunol. 2024 Jan 11;14:1330928. doi: 10.3389/fimmu.2023.1330928. eCollection 2023. PMID 38274807